CLINICAL TRIAL: NCT02832037
Title: A Phase II Randomised, Double-blinded, Placebo-controlled Parallel Group Trial to Examine the Efficacy and Safety of 4 Oral Doses of BI 425809 Once Daily Over 12 Week Treatment Period in Patients With Schizophrenia
Brief Title: Clinical Trial of BI 425809 Effect on Cognition and Functional Capacity in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1346.9; 2016-000285-28 (EudraCT Number)
Record Dates: First submitted 2016-07-07; First posted 2016-07-13 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

ARMS (5):
- BI 425809 dose 1 (Experimental)
  Interventions: Drug: BI 425809 dose 1; Drug: Placebo
- BI 425809 dose 2 (Experimental)
  Interventions: Drug: BI 425809 dose 2; Drug: Placebo
- BI 425809 dose 3 (Experimental)
  Interventions: Drug: BI 425809 dose 3; Drug: Placebo
- BI 425809 dose 4 (Experimental)
  Interventions: Drug: BI 425809 dose 4; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 425809 dose 1
  Arms: BI 425809 dose 1
Drug: BI 425809 dose 2
  Arms: BI 425809 dose 2
Drug: BI 425809 dose 3
  Arms: BI 425809 dose 3
Drug: BI 425809 dose 4
  Arms: BI 425809 dose 4
Drug: Placebo

SUMMARY:
The objective of the study is to investigate the efficacy, safety and pharmacokinetics of four different doses of BI 425809 once daily compared to placebo given for 12 weeks in patients with schizophrenia on stable antipsychotic treatment.

ELIGIBILITY:
Inclusion criteria:

* Men or women who are 18-50 years (inclusive) of age at time of consent
* Established schizophrenia with the following clinical features:

  * Outpatient, with no hospitalization for worsening of schizophrenia within 3 months prior to randomisation
  * Medically stable over the prior 4 weeks and psychiatrically stable without symptom exacerbation within 3 months prior to randomisation
  * patients who have no more than a moderate severe rating on the Positive and Negative Symptom Scale (PANSS) positive items P1, P3-P7 and no more than a moderate rating on the PANSS positive item P2
* Current antipsychotic and concomitant psychotropic medications as assessed at Visit 1 must meet the criteria below:

  * patients may have up to 2 antipsychotics (typical and/or atypical)
  * patients must be maintained on current typical and/or atypical antipsychotics other than Clozapine and on current dose for at least 4 weeks prior to randomisation and/or maintained on current long acting injectable antipsychotics and current dose for at least 3 months prior to randomization
  * patients must be maintained on current concomitant psychotropic medications, anticholinergics, antiepileptics and/or lithium for at least 3 months prior to randomisation and on current dose for at least 4 weeks prior to randomisation
* Women of child-bearing potential must be ready and able to use highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly.
* Patients must exhibit reliability, physiologic capability, and an educational level sufficient to comply with all protocol procedures, in the investigator´s opinion
* Patients must have an identified informant who will be consistent throughout the study.
* Further inclusion criteria apply

Exclusion criteria:

* Patients who have a categorical diagnosis of another current major psychiatric disorder
* Diseases of the central nervous system that may impact cognitive test performance
* Movement disorder not currently controlled
* Patients receiving another investigational drug or procedure within 30 days or 6 half-lives (whichever is longer) or recent participation in another trial with any cognitive enhancing therapy
* Recent participation in formal cognitive remediation program
* Recent electroconvulsive therapy
* Patients who have been on BI 409306, encenicline or other investigational drug testing effects on cognition in schizophrenia within the last 6 months prior to randomisation or who have previously been on bitopertin
* Participation in a clinical trial with repeated Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) assessments within the last 6 months
* Patients who required change in ongoing stable benzodiazepine or sleep medication regimen within the last 4 weeks prior to randomisation
* Treatment with Clozapine within 6 months prior to randomisation
* Treatment with medical devices (e.g. Transcranial Magnetic Stimulation (TMS), neurofeedback) for any psychiatric condition within the last 3 months prior to randomisation
* Patients taking strong or moderate Cytochrome P450 (CYPA4) inhibitors or inducers within the last 30 days prior to randomization
* Any suicidal behavior in the past 2 years (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior) prior to randomisation
* Any suicidal ideation of type 4 or 5 in the Columbia Suicidal Severity Rating Scale (C-SSRS) in the past 3 months (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent) prior to randomisation
* Known history of Human Immunodeficiency Virus (HIV) infection and/or a positive result for ongoing Hepatitis B or C infection on the Visit 1 central lab report
* Hemoglobin less than 120 g/L (12g/dL) in men or 115 g/L (11.5 g/dL) in women
* History of hemoglobinopathy such as thalassemia major or sickle-cell anemia
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial or men who are able to father a child, unwilling to be abstinent or use adequate contraception for the duration of the study participation and for at least 28 days after treatment has ended
* Significant history of drug abuse disorder (including alcohol) within the last 6 months prior to informed consent or a positive urine drug screen at screening (except for Benzodiazepines taken according to prescription and as an ongoing, stable regimen)
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 509 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (81):
- United States (21):
  - Collaborative Neuroscience Network, LLC (CNS), Garden Grove, California
  - Synergy San Diego, Lemon Grove, California
  - NRC Research Institute, Orange, California
  - Alliance for Wellness, Panorama City, California
  - CNRI - Los Angeles, Pico Rivera, California
  - CNRI-San Diego, LLC, San Diego, California
  - Premier Clinical Research Institute, Miami, Florida
  - Synexus, Atlanta, Georgia
  - Atlanta Center, Atlanta, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Lake Charles Clinical Trials LLC, Lake Charles, Louisiana
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - Mid-America Clinical Research, LLC, St Louis, Missouri
  - University at Buffalo, The State University of New York, Buffalo, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - North Carolina Psychiatric Research Center, Raleigh, North Carolina
  - Midwest Clinical Research, Dayton, Ohio
  - InSite Clinical Research, DeSoto, Texas
  - Psychiatric and Behavioral Solutions, LLC, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - AKH - Medical University of Vienna, Vienna
- Canada (5):
  - Dr. Alexander McIntyre Inc., Penticton, British Columbia
  - The Medical Arts Health Research Group, Vancouver, British Columbia
  - Chatham-Kent Clinical Trials Research Centre, Chatham, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
  - IUSMM Institut Universitaire en Sante Mentale de Montreal, Montreal, Quebec
- Germany (7):
  - Zentrum für klinische Forschung Dr. med. Irma Schöll & Kollegen, Bad Homburg
  - Praxis Dr. Volker Schumann, Berlin
  - Berufsausübungsgemeinschaft, Dr. sc. med. Alexander Schulze und Prof. Dr. med. Hagen Kunte, Berlin
  - Praxis Dr. Hahn, Berlin, Berlin
  - PANAKEIA Arzneimittelforschung Leipzig GmbH, Leipzig
  - Zentralinstitut für seelische Gesundheit, Mannheim
  - Neurologie und Psychiatrie / Psychotherapie, Westerstede
- Italy (3):
  - ASST degli Spedali Civili di Brescia, Concesio (BS)
  - Asst Santi Paolo E Carlo, Milan
  - Azienda Sanitaria Ospedale S. Luigi Gonzaga, Orbassano (TO)
- Japan (14):
  - Fujita Health University Hospital, Aichi, Toyoake
  - Chiba University Hospital, Chiba, Chiba
  - National Center for Global Health and Medicine Kohnodai Hospital, Chiba, Ichikawa
  - Hospital of the University of Occupational and Environmental Health, Fukuoka, Kitakyushu
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - Kobe University Hospital, Hyogo, Kobe
  - Kagawa University Hospital, Kagawa, Kita-gun
  - Kishiro Mental Clinic, Kanagawa, Kawasaki
  - Nara Medical University Hospital, Nara, Kashihara
  - Kansai Medical University Medical Center, Osaka, Moriguchi
  - Iwaki Clinic, Tokushima, Psychosomatic Medicine, Tokushima, Anan
  - National Center Neurology and Psychiatry, Tokyo, Kodaira
  - Showa University Karasuyama Hospital, Tokyo, Setagaya
  - Tokyo Women's Medical University Hospital, Tokyo, Shinjuku-ku
- Poland (7):
  - Wlokiennicza Med,Spec.Med.Prac,MD Tomasz Markowski,Bialystok, Bialystok
  - Podlassian Center of Psychogeriatry, Bialystok, Bialystok
  - Osrodek Badan Klinicznych CLINSANTE S.C., Bydgoszcz
  - Non-public Health Care Psychiatric Institution MENTIS,Leszno, Leszno
  - EUROMEDIS Sp. z o.o., Szczecin, Szczecin
  - Clin.Research Centre Clinsante SC Ewa Galczak-Nowak,Torun, Torun
  - Therapy Centre DIALOG Sp.z o.o. S.j., Warsaw
- South Korea (7):
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - National Center for Mental Health, Seoul
  - Asan Medical Center, Seoul
- Spain (6):
  - Hospital del Mar, Barcelona
  - Centro de Salud Mental de Fuencarral, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Puerta de Hierro, Majadahonda (Madrid)
  - Centro de Salud de San Juan, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
- Taiwan (4):
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei City Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (5):
  - Bushey Fields Hospital, Dudley
  - Royal Edinburgh Hospital, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - King's College Hospital, London
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Schultheis C, Rosenbrock H, Mack SR, Vinisko R, Schuelert N, Plano A, Sussmuth SD. Quantitative electroencephalography parameters as neurophysiological biomarkers of schizophrenia-related deficits: A Phase II substudy of patients treated with iclepertin (BI 425809). Transl Psychiatry. 2022 Aug 11;12(1):329. doi: 10.1038/s41398-022-02096-5. PMID 35953474
- [Derived] Fleischhacker WW, Podhorna J, Groschl M, Hake S, Zhao Y, Huang S, Keefe RSE, Desch M, Brenner R, Walling DP, Mantero-Atienza E, Nakagome K, Pollentier S. Efficacy and safety of the novel glycine transporter inhibitor BI 425809 once daily in patients with schizophrenia: a double-blind, randomised, placebo-controlled phase 2 study. Lancet Psychiatry. 2021 Mar;8(3):191-201. doi: 10.1016/S2215-0366(20)30513-7. PMID 33610228
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase II randomized, double-blind, double-dummy, placebo-controlled, multi-center, multi-national, 12-week parallel-group trial in participants with schizophrenia.
  Abbreviation: MMRM=Mixed-effects Model Repeated Measures
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 425809 2 mg Once a Day (q.d.): 2 milligram (mg) of BI 425809 administered orally (2 tablets with tablet strength 1 mg BI 425809, 1 placebo tablet matching 25 mg BI 425809 tablets) with water, with or without food, once daily in the morning. Continuous daily dosing for 12 weeks (planned treatment duration).
- BI 425809 5 mg q.d.: 5 milligram (mg) of BI 425809 administered orally (1 tablet with tablet strength 5 mg BI 425809, 1 placebo tablet matching 1 mg and 5 mg BI 425809 tablets, 1 placebo tablet matching 25 mg BI 425809 tablets) with water, with or without food, once daily in the morning. Continuous daily dosing for 12 weeks (planned treatment duration).
- BI 425809 10 mg q.d.: 10 milligram (mg) of BI 425809 administered orally (2 tablets with tablet strength 5 mg BI 425809, 1 placebo tablet matching 25 mg BI 425809 tablets) with water, with or without food in the morning, once daily. Continuous daily dosing for 12 weeks (planned treatment duration).
- BI 425809 25 mg q.d.: 25 milligram (mg) of BI 425809 administered orally (1 tablet with tablet strength 25 mg BI 425809, 2 placebo tablets matching 1 mg and 5 mg BI 425809 tablets) with water, with or without food, once daily in the morning. Continuous daily dosing for 12 weeks (planned treatment duration).
- Placebo q.d.: Placebo administered orally (2 placebo tablets matching 1 mg and 5 mg BI 425809 tablets, 1 placebo tablet matching 25 mg BI 425809 tablets) with water, with or without food, once daily in the morning. Continuous daily dosing for 12 weeks (planned treatment duration).
Period: Overall Study
Arm/Group | BI 425809 2 mg Once a Day (q.d.) | BI 425809 5 mg q.d. | BI 425809 10 mg q.d. | BI 425809 25 mg q.d. | Placebo q.d.
Started (= Randomized and Treated) | 85 | 84 | 85 | 85 | 170
Completed | 66 | 72 | 77 | 78 | 151
Not Completed | 19 | 12 | 8 | 7 | 19
Not completed — Administrative reasons | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 4 | 1 | 2
Not completed — Lost to Follow-up | 2 | 0 | 3 | 0 | 5
Not completed — Withdrawal by Subject | 9 | 8 | 0 | 4 | 8
Not completed — Adverse Event | 5 | 4 | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Population: The Treated Set included all participants who were randomized and were treated with at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 425809 2 mg Once a Day (q.d.) | BI 425809 5 mg q.d. | BI 425809 10 mg q.d. | BI 425809 25 mg q.d. | Placebo q.d. | Total
Number analyzed (Participants) | 85 | 84 | 85 | 85 | 170 | 509
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (8.5) | 37.5 (7.9) | 37.9 (6.8) | 36.2 (7.8) | 37.2 (7.7) | 37.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 27 | 24 | 35 | 60 | 180
  Male | 51 | 57 | 61 | 50 | 110 | 329
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 7 | 5 | 15 | 41
  Not Hispanic or Latino | 79 | 76 | 78 | 80 | 155 | 468
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 24 | 18 | 25 | 22 | 56 | 145
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 15 | 20 | 21 | 22 | 41 | 119
  White | 44 | 44 | 39 | 38 | 72 | 237
  More than one race | 2 | 1 | 0 | 2 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
MATRICS Consensus Cognitive Battery (MCCB) overall composite T-score [Mean (Standard Deviation); unit: Score on a scale] — The Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) overall composite T-score was derived from scores of seven cognitive domains (Speed of Processing, Verbal Learning, Working Memory, Reasoning and Problem Solving, Visual Learning, Social Cognition, Attention/Vigilance) obtained from a total of ten tests. MCCB overall composite T-score ranges typically between -20 and +99, where a larger MCCB overall composite T-score indicates better cognition.
  Score on a scale | 30.0 (13.8) | 32.8 (12.0) | 31.8 (12.8) | 30.2 (13.2) | 32.3 (13.6) | 31.5 (13.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cognitive Function as Measured by the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Overall Composite T-score After 12 Weeks of Treatment
Description: MCCB overall composite T-score was derived from scores of 7 cognitive domains (Speed of Processing, Verbal Learning, Working Memory, Reasoning and Problem Solving, Visual Learning, Social Cognition, Attention) obtained from a total of 10 tests (Trail Making, Brief Assessment of Cognition in Schizophrenia, Hopkins Verbal Learning, Wechsler Memory Scale, Letter-Number Span, Neuropsychological Assessment Battery, Brief Visuospatial Memory, Category Fluency, Mayer-Salovey-Caruso Emotional Intelligence, Continuous Performance) and ranges typically between -20 and +99, a larger T-score indicates better cognition.
  Change from baseline in MCCB overall composite T-score after 12 weeks of treatment was modeled using a MMRM with fixed, categorical factors of treatment at each visit, and continuous factors of baseline at each visit, using visit (week 6 and week 12 of treatment) as repeated measures, subject as random effect, adjusted mean (standard error) after 12 weeks of treatment is reported.
Time Frame: Baseline, after 6 and 12 weeks of treatment
Population: The Full Analysis Set included all participants who were randomized and were treated with at least 1 dose of trial medication and who had a non-missing baseline measurement and at least 1 non-missing post-baseline and on-treatment measurement for the primary or secondary efficacy endpoint.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | BI 425809 2 mg Once a Day (q.d.) | BI 425809 5 mg q.d. | BI 425809 10 mg q.d. | BI 425809 25 mg q.d. | Placebo q.d.
Number analyzed (Participants) | 79 | 80 | 82 | 83 | 163
scores on a scale | 1.784 (0.6805) | 1.641 (0.6656) | 3.486 (0.6410) | 3.234 (0.6410) | 1.504 (0.4579)
Statistical Analysis 1: Comparison: BI 425809 2 mg Once a Day (q.d.) vs BI 425809 5 mg q.d. vs BI 425809 10 mg q.d. vs BI 425809 25 mg q.d. vs Placebo q.d; A flat vs. non-flat dose-response relationship across the 4 doses of BI 425809 and placebo was tested using the Multiple Comparison Procedure - Modelling (MCP-Mod) approach which evaluated simultaneously 6 different plausible dose-response patterns (linear, linear in log, Emax, Sigmoid Emax, logistic, and beta) while protecting the overall probability of type I error (one-sided alpha of 0.05); Test type: Other — Mixed-effects Model Repeated Measures (MMRM) estimates were used as input for the MCP-Mod. MMRM included fixed, categorical factors of treatment, analysis visit as repeated measures per subject, and treatment by analysis visit interaction, continuous fixed covariate of baseline value and baseline value by analysis visit interaction, subject as random effect, covariance structure= Unstructured; p = 0.0145, MCP-Mod linear model fit — Adjusted for multiplicity
Statistical Analysis 2: Comparison: BI 425809 2 mg Once a Day (q.d.) vs BI 425809 5 mg q.d. vs BI 425809 10 mg q.d. vs BI 425809 25 mg q.d. vs Placebo q.d; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0148, MCP-Mod linear in log model fit — Adjusted for multiplicity
Statistical Analysis 3: Comparison: BI 425809 2 mg Once a Day (q.d.) vs BI 425809 5 mg q.d. vs BI 425809 10 mg q.d. vs BI 425809 25 mg q.d. vs Placebo q.d; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0089, MCP-Mod Emax model fit — Adjusted for multiplicity; Model assumption: 20% of the maximum effect is achieved at 2 mg of BI 425809
Statistical Analysis 4: Comparison: BI 425809 2 mg Once a Day (q.d.) vs BI 425809 5 mg q.d. vs BI 425809 10 mg q.d. vs BI 425809 25 mg q.d. vs Placebo q.d; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0038, MCP-Mod Sigmoid Emax model fit — Adjusted for multiplicity; Model assumption: 25% of the maximum effect is achieved at 5 mg and 75% of the maximum effect is achieved at 10 mg of BI 425809
Statistical Analysis 5: Comparison: BI 425809 2 mg Once a Day (q.d.) vs BI 425809 5 mg q.d. vs BI 425809 10 mg q.d. vs BI 425809 25 mg q.d. vs Placebo q.d; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0085, MCP-Mod logistic model fit — Adjusted for multiplicity; Model assumption: 10% of the maximum effect is achieved at 5 mg and 50% of the maximum effect is achieved at 10 mg of BI 425809
Statistical Analysis 6: Comparison: BI 425809 2 mg Once a Day (q.d.) vs BI 425809 5 mg q.d. vs BI 425809 10 mg q.d. vs BI 425809 25 mg q.d. vs Placebo q.d; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2280, MCP-Mod beta model fit — Adjusted for multiplicity; Assumption:75% of maximum (max) effect at 2mg, 87.5% of max effect at 5mg,25% of max effect at 25mg,max effect at 10mg BI 425809, scalar parameter=26
Statistical Analysis 7: Comparison: BI 425809 2 mg Once a Day (q.d.) vs Placebo q.d; Secondary analysis. No formal hypotheses were tested; Test type: Other — Mixed Model Repeated Measures included fixed, categorical factors of treatment, analysis visit as repeated measures per subject, and treatment by analysis visit interaction, continuous fixed covariate of baseline value and baseline value by analysis visit interaction, subject as random effect, covariance structure= Unstructured; p = 0.7330, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = 0.280, 95% CI 2-sided [-1.332 to 1.892], Standard Error of Mean 0.8205 — Difference was calculated as BI 425809 - placebo
Statistical Analysis 8: Comparison: BI 425809 5 mg q.d. vs Placebo q.d; Secondary analysis. No formal hypotheses were tested; Test type: Other — [test comment as in outcome 1, analysis 7]; p = 0.8655, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = 0.137, 95% CI 2-sided [-1.450 to 1.724], Standard Error of Mean 0.8074 — Difference was calculated as BI 425809 - placebo
Statistical Analysis 9: Comparison: BI 425809 10 mg q.d. vs Placebo q.d; Secondary analysis. No formal hypotheses were tested; Test type: Other — [test comment as in outcome 1, analysis 7]; p = 0.0122, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = 1.982, 95% CI 2-sided [0.434 to 3.530], Standard Error of Mean 0.7875 — Difference was calculated as BI 425809 - placebo
Statistical Analysis 10: Comparison: BI 425809 25 mg q.d. vs Placebo q.d; Secondary analysis. No formal hypotheses were tested; Test type: Other — [test comment as in outcome 1, analysis 7]; p = 0.0287, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = 1.730, 95% CI 2-sided [0.181 to 3.280], Standard Error of Mean 0.7884 — Difference was calculated as BI 425809 - placebo

2. Secondary Outcome: Change From Baseline in Everyday Functional Capacity as Measured by Schizophrenia Cognition Rating Scale (SCoRS) Total Score After 12 Weeks of Treatment
Description: SCoRS total score was derived as the sum of non-missing responses from 20 interview-based items rated by an interviewer on a 4-point scale. A response of "not available" to an item was treated as missing. If six or more of the 20 items were missing for a participant at a visit, then the corresponding SCoRS total score was missing for that participant at the visit. If five or less of the 20 items were missing for a participant at a visit, then the item(s) with missing value(s) were imputed first with the average of the non-missing item values, then the SCoRS total score for the participant at the visit was derived as the sum of non-missing item values and the imputed item values. SCoRS total score is between 20 and 80 where higher score values represent greater degree of impairment in day-to-day functions due to cognitive deficits.
  Analysis of covariance model was fitted to calculate adjusted mean and standard error, model details in the Statistical Analysis section.
Time Frame: Baseline and after 12 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BI 425809 2 mg Once a Day (q.d.) | BI 425809 5 mg q.d. | BI 425809 10 mg q.d. | BI 425809 25 mg q.d. | Placebo q.d.
Number analyzed (Participants) | 77 | 80 | 82 | 83 | 158
units on a scale | -1.637 (0.5992) | -3.652 (0.5890) | -3.078 (0.5803) | -3.887 (0.5770) | -2.815 (0.4181)
Statistical Analysis 1: Comparison: BI 425809 2 mg Once a Day (q.d.) vs BI 425809 5 mg q.d. vs BI 425809 10 mg q.d. vs BI 425809 25 mg q.d. vs Placebo q.d; [analysis description as in outcome 1, analysis 1]; Test type: Other — Analysis of covariance (ANCOVA) model estimates were used as input for the MCP-Mod. ANCOVA included treatment as fixed categorical factor, and baseline score as continuous fixed covariate; p = 0.0660, MCP-Mod linear model fit — P-value is considered nominal
Statistical Analysis 2: Comparison: BI 425809 2 mg Once a Day (q.d.) vs BI 425809 5 mg q.d. vs BI 425809 10 mg q.d. vs BI 425809 25 mg q.d. vs Placebo q.d; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.1619, MCP-Mod linear in log model fit — P-value is considered nominal
Statistical Analysis 3: Comparison: BI 425809 2 mg Once a Day (q.d.) vs BI 425809 5 mg q.d. vs BI 425809 10 mg q.d. vs BI 425809 25 mg q.d. vs Placebo q.d; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0832, MCP-Mod Emax model fit — P-value is considered nominal; Model assumption: 20% of the maximum effect is achieved at 2 mg of BI 425809
Statistical Analysis 4: Comparison: BI 425809 2 mg Once a Day (q.d.) vs BI 425809 5 mg q.d. vs BI 425809 10 mg q.d. vs BI 425809 25 mg q.d. vs Placebo q.d; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0625, MCP-Mod Sigmoid Emax model fit — P-value is considered nominal; [statistical method as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: BI 425809 2 mg Once a Day (q.d.) vs BI 425809 5 mg q.d. vs BI 425809 10 mg q.d. vs BI 425809 25 mg q.d. vs Placebo q.d; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0768, MCP-Mod logistic model fit — P-value is considered nominal; [statistical method as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: BI 425809 2 mg Once a Day (q.d.) vs BI 425809 5 mg q.d. vs BI 425809 10 mg q.d. vs BI 425809 25 mg q.d. vs Placebo q.d; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.7479, MCP-Mod beta model fit — P-value is considered nominal; [statistical method as in outcome 1, analysis 6]
Statistical Analysis 7: Comparison: BI 425809 2 mg Once a Day (q.d.) vs Placebo q.d; Secondary analysis. No formal hypotheses were tested; Test type: Other; p = 0.11, ANCOVA — P-value is considered nominal; Analysis of covariance (ANCOVA) model included treatment as fixed categorical factor, and baseline score as continuous fixed covariate; Difference of adjusted means = 1.178, 95% CI 2-sided [-0.258 to 2.613], Standard Error of Mean 0.7306 — Difference was calculated as BI 425809 - placebo
Statistical Analysis 8: Comparison: BI 425809 5 mg q.d. vs Placebo q.d; Secondary analysis. No formal hypotheses were tested; Test type: Other; p = 0.25, ANCOVA — P-value is considered nominal; [statistical method as in outcome 2, analysis 7]; Difference of adjusted means = -0.837, 95% CI 2-sided [-2.257 to 0.582], Standard Error of Mean 0.7224 — Difference was calculated as BI 425809 - placebo
Statistical Analysis 9: Comparison: BI 425809 10 mg q.d. vs Placebo q.d; Secondary analysis. No formal hypotheses were tested; Test type: Other; p = 0.71, ANCOVA — P-value is considered nominal; [statistical method as in outcome 2, analysis 7]; Difference of adjusted means = -0.263, 95% CI 2-sided [-1.669 to 1.142], Standard Error of Mean 0.7152 — Difference was calculated as BI 425809 - placebo
Statistical Analysis 10: Comparison: BI 425809 25 mg q.d. vs Placebo q.d; Secondary analysis. No formal hypotheses were tested; Test type: Other; p = 0.13, ANCOVA — P-value is considered nominal; [statistical method as in outcome 2, analysis 7]; Difference of adjusted means = -1.072, 95% CI 2-sided [-2.473 to 0.328], Standard Error of Mean 0.7125 — Difference was calculated as BI 425809 - placebo

3. Secondary Outcome: Percentage of Participants With Any Adverse Event
Description: Percentage of participants with any Adverse Event.
Time Frame: On-treatment period, that is, from first intake of any trial drug until the last intake of any trial drug (planned: 84 days) + residual effect period (11 days), up to 103 days
Population: The Treated Set included all participants who were randomized and were treated with at least 1 dose of trial medication.
Measure: Number; unit: Percentage of participants
Arm/Group | BI 425809 2 mg Once a Day (q.d.) | BI 425809 5 mg q.d. | BI 425809 10 mg q.d. | BI 425809 25 mg q.d. | Placebo q.d.
Number analyzed (Participants) | 85 | 84 | 85 | 85 | 170
Percentage of participants | 58.8 | 52.4 | 41.2 | 42.4 | 43.5

ADVERSE EVENTS:
Time Frame: For Serious and Other Adverse Events: On-treatment period, that is, from first intake of any trial drug until the last intake of any trial drug (planned: 84 days) + residual effect period (11 days), up to 103 days. For All-Cause Mortality: On-treatment period + Follow-up period (planned: 28±7 days), up to 127 days.
Description: The Treated Set included all participants who were randomized and were treated with at least 1 dose of trial medication.
Arm/Group | BI 425809 2 mg Once a Day (q.d.) | BI 425809 5 mg q.d. | BI 425809 10 mg q.d. | BI 425809 25 mg q.d. | Placebo q.d.
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/84 | 0/85 | 0/85 | 0/170
Serious Adverse Events (participants affected / at risk) | 2/85 | 4/84 | 2/85 | 4/85 | 4/170
Other Adverse Events (participants affected / at risk) | 22/85 | 23/84 | 14/85 | 13/85 | 31/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 425809 2 mg Once a Day (q.d.) (N=85) | BI 425809 5 mg q.d. (N=84) | BI 425809 10 mg q.d. (N=85) | BI 425809 25 mg q.d. (N=85) | Placebo q.d. (N=170)
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infective myositis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Drug dependence (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Fear of disease (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Psychotic symptom (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 425809 2 mg Once a Day (q.d.) (N=85) | BI 425809 5 mg q.d. (N=84) | BI 425809 10 mg q.d. (N=85) | BI 425809 25 mg q.d. (N=85) | Placebo q.d. (N=170)
Nasopharyngitis (Infections and infestations) | 8 | 9 | 7 | 4 | 13
Dizziness (Nervous system disorders) | 5 | 4 | 2 | 3 | 6
Headache (Nervous system disorders) | 8 | 10 | 7 | 8 | 9
Somnolence (Nervous system disorders) | 2 | 5 | 5 | 2 | 4

LIMITATIONS AND CAVEATS:
After identifying a new major metabolite (BI 761036), the sponsor communicated a voluntary hold of Phase II to relevant competent authorities on 16-Sep-2016. This was formalized to a full clinical hold of the development program by the Food and Drug Administration (FDA) on 26-Oct-2016. Before start of the hold, 1 patient was screened, but not randomized. Clinical hold was removed by FDA on 21-Nov-2017, the trial was re-initiated with version 3 of the clinical trial protocol, dated 13-Dec-2017.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT02832037/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT02832037/SAP_001.pdf